CLINICAL TRIAL: NCT04733144
Title: An Bioequivalence Study of Prednisolone and Dexamethasone; Corticosteroids Revised - The CORE Study
Brief Title: Bioequivalence Study of Prednisolone and Dexamethasone
Acronym: CORE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, A.P. van Beek, MD PhD, Dr. A.P. van Beek, Endocrinologist, Principal Investigator, University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 201900874; 2019-004983-23 (EudraCT Number)
Record Dates: First submitted 2021-01-15; First posted 2021-02-01 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Prednisolone; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisolone-Dexamethasone (Active Comparator): Participants will receive 1 week of low dose (7,5 mg) prednisolone directly followed by 1 week of high dose prednisolone (30 mg). After a wash-out period, participants in this arm will receive 1 week of low dose dexamethasone (1,125 mg) directly followed by 1 week of high dose dexamethasone (4,5 mg).
  Interventions: Drug: Prednisolone; Drug: Dexamethasone
- Dexamethasone-Prednisolone (Active Comparator): Participants will receive 1 week of low dose (1,125 mg) dexamethasone directly followed by 1 week of high dose dexamethasone (30 mg). After a wash-out period, participants in this arm will receive 1 week of low dose prednisolone (7,5 mg) directly followed by 1 week of high dose prednisolone (30 mg).
  Interventions: Drug: Prednisolone; Drug: Dexamethasone

INTERVENTIONS:
Drug: Prednisolone — 7,5 mg prednisolone (low dose) 30 mg prednisolone (high dose)
Drug: Dexamethasone — 1,125 mg dexamethasone 4,5 mg dexamethasone

SUMMARY:
The purpose of this study is to compare two different glucocorticoids, prednisolone and dexamethasone at two different doses for their organ specific effects, utilizing modern day standards.

DETAILED DESCRIPTION:
Study design: A randomised, double blind, cross-over clinical trial.

Study population: healthy human adult volunteers including 12 males and 12 females aged 18-75 years old.

Intervention: In random order, subjects will receive 7,5 mg prednisolone for one week, directly followed by 30 mg of prednisolone for one week. After a washout period of 4 weeks (or by exception 8 weeks), subjects will receive 1,125 mg dexamethasone for one week, directly followed by 4,5 mg dexamethasone for one week.

Main study parameters/endpoints: The main study endpoint is the difference in total urinary cortisol excretion as measured in 24h-urine between the lower doses of prednisolone and dexamethasone as well as between the higher doses of prednisolone and dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy with no relevant medical history and no use of medication.
* Female participants aged <50 years must be using oral contraceptives and female participants age ≥50 years must be in the postmenopausal state
* Command of the Dutch language
* Providing written IC
* BMI between 18.5 and 30 kg/m2
* Participants must be between 18 and 75 years of age

Exclusion Criteria:

* Potential participants who are unlikely to adhere to the study protocol (for instance subjects which have a history of substance abuse or non-compliance)
* Potential participants with a medical history of:

  1. Diseases affecting the HPA-axis: e.g. primary and secondary adrenal insufficiency, pituitary tumors, and nightshift workers
  2. Diseases affecting the HPG-axis: e.g. Cushing disease.
  3. Chronic inflammatory diseases: e.g. rheumatoid arthritis, polymyalgia rheumatic, and asthma
  4. Psychiatric diseases
  5. Diabetes
* Shift workers
* Potential participants with a kidney function <60 ml/min/1.73m2, abnormalities in liver enzymes, and/or abnormalities in thyroid function
* Potential participants who are dependent on corticosteroids, e.g. asthmatic patients, and transplant recipients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Suppression of the hypothalamic-pituitary-adrenal axis - low dose | 1 week per treatment
  Difference in HPA-axis suppression as measured by the difference of total urinary cortisol excretion in 24h-urine between 7,5 mg prednisolone and 1,125 mg dexamethasone
Suppression of the hypothalamic-pituitary-adrenal axis - high dose | 1 week per treatment
  Difference of total urinary cortisol excretion in 24h-urine between 30 mg prednisolone (preceded by 7,5 mg prednisolone for one week) and 4,5 mg dexamethasone (preceded by 1,125 mg dexamethasone for one week)

SECONDARY OUTCOMES:
Changes in hypothalamic-pituitary-adrenal axis suppression - 1 | 1 week per treatment
  Effect of a dosage increase from low dose to high dose prednisolone on total urinary cortisol excretion in 24h-urine
Changes in hypothalamic-pituitary-adrenal axis suppression - 2 | 1 week per treatment
  Effect of a dosage increase from low dose to high dose dexamethasone on total urinary cortisol excretion in 24h-urine
Suppression of the hypothalamic-pituitary-adrenal axis - plasma cortisol | 1 week per treatment
  The between-group difference in plasma cortisol levels
Suppression of the hypothalamic-pituitary-adrenal axis - ACTH | 1 week per treatment
  The between-group difference in adrenocorticotropic hormone levels
Suppression of the hypothalamic-pituitary-adrenal axis - metabolites of the 24h-urine steroid profile | 1 week per treatment
  The between-group difference in metabolites of the 24h-urine steroid profile
Suppression of the hypothalamic-pituitary-gonadal axis - androgen profile | 1 week per treatment
  The between-group difference in androgen profiles
Suppression of the hypothalamic-pituitary-gonadal axis - gonadotropins | 1 week per treatment
  The between-group difference in luteinizing hormone and follicle stimulating hormone
Suppression of the hypothalamic-pituitary-gonadal axis - metabolites of the 24h-urine steroid profile | 1 week per treatment
  The between-group difference in metabolites of the 24h-urine steroid profile
Pharmacokinetics | 1 week per treatment
  Area under the curve
Suppression of the immune system - granulocyte count | 1 week per treatment
  The between-group difference in granulocyte count
Suppression of the immune system - PBMCs | 1 week per treatment
  The between-group difference in peripheral blood mononuclear cell count
Effect on blood pressure | 1 week per treatment
  The between-group difference in systolic and diastolic blood pressure
Effect on the Renin-angiotensin-aldosterone system - plasma renin | 1 week per treatment
  The between-group difference in plasma renin
Effect on the Renin-angiotensin-aldosterone system - aldosterone | 1 week per treatment
  The between-group difference in aldosterone
Effect on the Renin-angiotensin-aldosterone system - plasma potassium | 1 week per treatment
  The between-group difference in plasma potassium
Effect on the Renin-angiotensin-aldosterone system - 24h-urine potassium | 1 week per treatment
  The between-group difference in 24h-urine potassium
Effect on the Renin-angiotensin-aldosterone system - trans-tubular potassium gradient | 1 week per treatment
  The between-group difference in trans-tubular potassium gradient
Metabolic parameters - OGTT | 1 week per treatment
  The between-group difference in oral glucose tolerence tests
Metabolic parameters - lipid profile | 1 week per treatment
  The between-group difference in lipid profile
Metabolic parameters - NEFAs | 1 week per treatment
  The between-group difference in non-esterified fatty acids
Muscle mass | 1 week per treatment
  The between-group difference in 24h urinary creatinine excretion rate
Muscle strength | 1 week per treatment
  The between-group difference in handgrip strength
Clinical parameters - Weight | 1 week per treatment
  The between-group difference in weight in kg
Clinical parameters - Body Mass Index (BMI) | 1 week per treatment
  The between-group difference in BMI in kg/m2
Clinical parameters - Waist circumference | 1 week per treatment
  The between-group difference in waist circumference in cm
Clinical parameters - Hip circumference | 1 week per treatment
  The between-group difference in hip circumference in cm
Questionnaires - Quality of life | 1 week per treatment
  The between-group difference in quality of life, measured using the 36-Item Short Form Health Survey (SF-36). The score ranges from 0-100, with lower scores indicating a worse health status.
(Serious) Adverse Events | 1 week per treatment
  The between-group difference in (serious) adverce events

CONTACTS AND LOCATIONS:
Overall Officials: André P. van Beek, MD,PhD, Principal Investigator — University Medical Center Groningen; Stephan J.L. Bakker, MD,PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
After deidentification, individual data that are the foundation of the results reported in future manuscripts can be made available (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 6 months and ending 10 years following article publication
Access Criteria: Researchers should provide a methodologically sound proposal to a.p.van.beek@umcg.nl

REFERENCES:
- [Derived] Stam SP, Vulto A, Vos MJ, Kerstens MN, Rutgers A, Kema I, Touw DJ, Bakker SJ, van Beek AP. Rationale and design of the CORE (COrticosteroids REvised) study: protocol. BMJ Open. 2022 Apr 26;12(4):e061678. doi: 10.1136/bmjopen-2022-061678. PMID 35473729